CLINICAL TRIAL: NCT00507962
Title: A Phase I Study Dose Escalation Clinical Study Of Hepatic Intraarterial Cisplatin, In Combination With Systemic Intravenous Liposomal Doxorubicin Administered Every Four Weeks to Patients With Advanced Cancer And Dominant Liver Involvement
Brief Title: Cisplatin HAI Study in Patients With Advanced Cancer and Dominant Liver Involvement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0568
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Dominant Liver Involvement; Hepatic Intraarterial Cisplatin; Cisplatin; Liposomal Doxorubicin; Platinol-AQ; Platinol; CDDP; Doxil; Liposomal; Doxorubicin Hydrochloride
MeSH Terms: interventions — Cisplatin; liposomal doxorubicin; Liposomes; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin + Liposomal Doxorubicin (Experimental): Cisplatin 100 mg/m^2 Intraarterial and Liposomal Doxorubicin starting dose 20 mg/m^2 by vein on Day 1 every 4 weeks
  Interventions: Drug: Cisplatin; Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: Cisplatin — 100 mg/m^2 Intraarterial On Day 1 Every 4 Weeks
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Liposomal Doxorubicin — Starting dose 20 mg/m^2 IV On Day 1 Every 4 Weeks
  Other Names: Doxil; Liposomal; Doxorubicin Hydrochloride

SUMMARY:
The goal of this clinical research study is find the highest safe dose of cisplatin that can be given with liposomal doxorubicin in the treatment of advanced cancer involving the liver.

PRIMARY Objectives:

To determine the toxicity and safety of a monthly cytotoxic regimen combining intraarterial hepatic (HAI) cisplatin with systemic intravenous liposomal doxorubicin in patients with cancer metastatic to the liver.

SECONDARY Objectives:

To document in a descriptive fashion the antitumor efficacy of monthly hepatic intraarterial cisplatin in combination with systemic liposomal doxorubicin.

DETAILED DESCRIPTION:
Cisplatin and Liposomal Doxorubicin are chemotherapy drugs designed to fight cancer growth.

If you are eligible to take part in this study, you will enter a treatment period that is divided into cycles. Each cycle is 28 days. You will be hospitalized to receive your chemotherapy. The night of the hospital admission you will receive fluids (normal saline) in your veins to help avoid kidney side effects from the chemotherapy. The morning after your admission to the hospital you will be taken to the interventional radiology suite and a catheter will be placed in your right groin. You must be on bedrest the entire time that the catheter is in place. After the procedure, you will go to Nuclear Medicine and a test called "flow study" will be carried out to confirm the right position of the catheter. After your return to the room, the nurses will start the chemotherapy. You will first receive cisplatin through the groin catheter followed by the liposomal doxorubicin given in one of your veins. The treatment lasts less than three hours and is repeated once every month.

The catheter will be carefully taped so it can not move and to prevent it from coming out. Following completion of chemotherapy infusion, the intra-arterial catheter will be pulled and pressure applied to the groin for 15 minutes. In some cases, the catheter will be removed immediately after your chemotherapy infusions is complete. In some cases, the catheter will remain in longer. You will be on bedrest until the catheter is removed. The catheter will be removed by the physician on call. The catheter will be placed and removed at each treatment.

Blood (about 2 teaspoons) will be drawn for blood counts and liver function tests before each dose to be sure researchers are safely giving you the liposomal doxorubicin.

Since most of the blood flow to your liver comes through the portal vein, your doctors will try to cause an infarct (like a stroke) to the liver artery followed by the injection of cisplatin to kill the tumor cells.

You will be seen by a doctor or advanced practice practitioner every day while you are in the hospital. You will be hospitalized for about 5-7 days until recovery from all immediate treatment related side effects.

You will continue to receive therapy as mentioned above until the disease gets worse or intolerable side effects occur.

At the end of your participation in this study, you will have scans to see if your tumors are growing or shrinking, and blood work (about 3 teaspoons) to make sure your blood counts and the electrolytes (salts in your blood), kidney and liver function are at a safe level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Histologically confirmed diagnosis of malignancy and liver involvement as dominant site of metastasis (over 50% of all tumor burden).
2. Pediatric patients eligible at the discretion of the primary investigator.
3. Performance Status Equivalent or Grater than 60% in the Karnofsky's Performance scale (Requires occasional assistance but is able to care for own needs).
4. Adequate Renal Function (Serum CRE </= 1.5 mg/dL) or calculated Creatinine Clearance >/= 50 ml/min (Cockcroft Formula).
5. Adequate Hepatic Function (Total Bilirubin </= 1.5 mg/dL or ALT </= 5 times upper normal reference value).
6. Adequate Bone Marrow Function (Absolute neutrophil count (ANC) >/= 1.5 cells/uL; number of platelets (PLT) >/= 100,000 cells/uL).
7. At least three weeks from previous cytotoxic chemotherapy before day 1 of HAI infusion. After targeted or biologic therapy there should be 5 half-lives or three weeks, whichever is shorter.
8. All Females in Childbearing Age MUST have a negative urine or serum Human chorionic gonadotropin or human chorionic gonadotrophin (hCG) test unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity).
9. Ability to fully read, comprehend, and sign informed consent forms. In pediatric patients, the informed consent forms will be signed by a parent or legal guardian.
10. Patients with germ cell tumors and lymphoma MUST have had documented progression of disease prior to enrollment.

Exclusion Criteria:

1. Clinical or radiographic evidence of Ascites.
2. Pregnant females.
3. Hypersensitivity to platinum compounds or anthracyclines.
4. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
5. Jaundice. (Bilirubin > 1.5 mg/dL).
6. Bleeding Diathesis.(Prothrombin time > 20 secs or International Normalized Ratio (INR) > 2.0).
7. Portal vein thrombosis.
8. Grade 2 Peripheral Neuropathy (CTC V3.0: Sensory alteration interfering with function but not interfering with ADL)
9. Medical History or Clinical Evidence of Congestive Heart Failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | With each 4 week cycle (28 days)
  Dose level at which no dose limiting toxicities are seen for a monthly cytotoxic regimen combining intraarterial hepatic cisplatin with systemic intravenous liposomal doxorubicin.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org